CLINICAL TRIAL: NCT05149846
Title: Effect of Pre-conditioning by Balloon-inflation on Myocardial Injury During Complex Percutaneous Coronary Intervention - a Clinical Trial
Brief Title: Pre-conditioning by Balloon-inflation on Myocardial Injury
Acronym: BaMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BaMI
Record Dates: First submitted 2021-11-11; First posted 2021-12-08 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2021-11

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-conditioning (Other): Pre-conditioning by three consecutive 60 seconds balloon inflations, spaced 120 seconds apart followed by 10 minutes rest prior to PCI
  Interventions: Procedure: Pre-conditioning
- Controll (No Intervention): No pre-conditioning, standard care

INTERVENTIONS:
Procedure: Pre-conditioning — Pre-conditioning by three consecutive 60 seconds balloon inflations, spaced 120 seconds apart followed by 10 minutes rest prior to PCI
  Arms: Pre-conditioning

SUMMARY:
Study objectives:

To test pre-conditioning by three consecutive 60 seconds balloon inflations, spaced 120 seconds apart, followed by 10 minutes rest prior to PCI reduces the risk of myocardial injury.

Study design:

Single-center, open-label, randomized controlled trial

Study population:

Patients with indication for complex PCI. Patients will be randomized prior to PCI to pre-conditioning by intracoronary balloon inflation in the target vessel proximal to the target lesion(s) versus no pre-conditioning followed by a 10-minute waiting period prior to PCI. PCI will then be performed as per standard of care. Cardiac biomarkers will be drawn at baseline and 6, 24 and 48 hours after PCI. Cardiac magnetic resonance imaging will be performed at 48 hours and 6 months post PCI.

DETAILED DESCRIPTION:
The primary objective of this study is to test pre-conditioning by three consecutive 60 seconds balloon inflations, spaced 120 seconds apart followed by 10 minutes rest prior to percutaneous coronary intervention (PCI) reduces the risk of myocardial injury.

Except for the extended duration of balloon inflations, no study-specific therapy will be administered to the patients. All patients will receive treatment according to current guidelines. A follow-up visit will be performed at approximately 6, 24, 48 hours and at 6 months.

The population studied are patients with indication for complex PCI. Patients will be randomized, after providing written informed consent, prior to PCI to pre-conditioning by three consecutive intracoronary balloon inflation in the target vessel proximal to the target lesion(s) versus no pre-conditioning followed by a 10-minute waiting period prior to PCI, PCI will then be performed as per standard of care. Cardiac biomarkers will be drawn at baseline and 6 hours, 24 hours and 48 hours after PCI. Cardiac magnetic resonance imaging will be performed at 48 hours and 6 months post PCI.

Three consecutive balloon occlusions performed for approximate 60 seconds and spaced approximate 120 seconds apart, followed by a 10-minute waiting period prior to PCI.

Cardiac Magnetic Resonance imaging (CMR) will be used to assess size of myocardial infarction at 48±6 hours and 6 months±30 days post PCI. CMR examination includes administration of contrast and one additional blood test (hematocrit, necessary to assess extracellular volume).

Echocardiography can be used before randomization as per standard of care before PCI. Echocardiography will be used to assess wall motion score index, left ventricular ejection fraction at 24 hours and serial examinations can be performed at the discretion of the PI 12-lead Electrocardiogram (ECG) will be used to assess at baseline, during intervention, at 48 hours and serial examinations can be performed at the discretion of the PI.

Apart from the routine laboratory tests, blood samples (troponin-I, troponin-T, creatine kinase MB fraction [CKMB]) will be collected at baseline, 6±1 hour, 24±6 hours 48±6 hours after PCI. After collection blood samples will be analyzed at hospitals clinical laboratory and destructed directly after analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Indication for complex PCI, defined as:

   1. PCI of a chronic total occlusion
   2. Two-stent PCI of a bifurcation lesion.
   3. PCI of severely calcified lesion
3. Preprocedural biomarker Troponin-I within normal range
4. Left ventricular ejection fraction >50%
5. Written informed consent obtained

Exclusion Criteria:

1. Previous randomization in the study
2. Decompensated heart failure requiring inotropic /adrenergic support, invasive or non-invasive ventilation or intra-aortic balloon pump/ventricular assist device therapy less than 48 hours prior to randomization
3. Recent PCI (<3 months)
4. Known previous myocardial infarction in the target vessel or regional wall motion abnormalities within the myocardium subtended by the target vessel(s)
5. Any contraindication for Cardiac magnetic resonance imaging
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac troponin-I | within 48 hours
  Area-under the curve of cardiac troponin-I
Infarct size | 48 hours
  Procedural infarct size as assessed by cardiac magnetic resonance imaging
Infarct size | 6 months
  Procedural infarct size as assessed by cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Björn Redfors, MD, PhD, Principal Investigator — Vastra Gotaland Region